CLINICAL TRIAL: NCT02620774
Title: Tissue Penetration of Ceftolozane/Tazobactam in Diabetic Patients With Lower Limb Infections
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hartford Hospital (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: Nicolau-53433
Record Dates: First submitted 2015-12-01; First posted 2015-12-03 (Estimated); Results first posted 2019-01-15 (Actual); Last update posted 2019-01-15 (Actual); Status verified 2017-10

CONDITIONS: Diabetes; Wound Infection; Healthy Volunteers
MeSH Terms: conditions — Diabetes Mellitus; Wound Infection | interventions — ceftolozane, tazobactam drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Diabetic Wound Infection (Experimental): Participants with a documented history of Type 1 or Type 2 diabetes and a mild to moderate (Grade 2 or 3) wound infection of the lower limb will receive at least 3 doses of intravenous ceftolozane/tazobactam 1.5g every 8 hours, followed by sampling of interstitial tissue fluid at the margin of the wound by a microdialysis probe over 8 hours.
  Interventions: Drug: Ceftolozane/tazobactam; Procedure: Microdialysis Catheter Insertion
- Healthy Volunteer (Active Comparator): Participants will be male or female healthy adult volunteers with no significant medical or medication history. Participants will receive at least 3 doses of intravenous ceftolozane/tazobactam 1.5g every 8 hours, followed by sampling of interstitial tissue fluid in the thigh by a microdialysis probe over 8 hours.
  Interventions: Drug: Ceftolozane/tazobactam; Procedure: Microdialysis Catheter Insertion

INTERVENTIONS:
Drug: Ceftolozane/tazobactam — 3 or more doses of ceftolozane/tazobactam intravenously administered over 60 minutes every 8 hours
  Other Names: Zerbaxa
Procedure: Microdialysis Catheter Insertion — A 20 kila-Dalton microdialysis probe (63 MD catheter; MDialysis Inc., N. Chelmsford, MA) will be inserted into the subcutaneous tissue at the margin of the wound (patient group) or in the thigh tissue (healthy volunteers). The probe will be left in place for the final dose and all tissue sampling procedures thereafter. This probe is perfused with a physiologic solution to collect interstitial fluid samples. The probe will then be removed after completion of sample collection.

SUMMARY:
This study will determine the tissue penetration of ceftolozane/tazobactam (Zerbaxa, Merck & Co.), a novel β-lactam/β-lactamase combination antibiotic, into the extracellular, interstitial fluid of soft tissue in diabetic patients with lower limb wound infections. Penetration will be compared with a group of healthy volunteer control participants.

DETAILED DESCRIPTION:
This study will enroll 10 patients with diabetes who are admitted with a lower limb wound infection and 6 healthy volunteer control participants. The study will take place in an inpatient unit at Hartford Hospital for all patients and in the Clinical Research Center at Hartford Hospital for all healthy volunteers. All participants will receive at least 3 doses of ceftolozane/tazobactam 1.5g every 8 hours. A microdialysis probe (Mdialysis Inc., N. Chelmsford MA) will be inserted into the subcutaneous soft tissue near the margin of the wound (patients) or in the thigh (healthy volunteers). The microdialysis probe is perfused with lactated Ringer's solution and samples are collected each hour for 8 hours after the final dose. A peripheral intravenous catheter will be inserted into an arm vein to collect blood samples simultaneously with microdialysis samples. Concentrations in tissue are compared with blood to determine percent penetration.

ELIGIBILITY:
Inclusion Criteria:

* Experimental: Type 1 or Type 2 diabetes and a mild to moderate (Grade 2 or 3) wound infection of the lower limb
* Active Comparator: Healthy Adult Volunteer

Exclusion Criteria:

All Participants:

* Less than 18 years of age
* History of hypersensitivity to ceftolozane/tazobactam, piperacillin/tazobactam, or any β-lactam antibiotic
* History of hypersensitivity to lidocaine or lidocaine derivatives
* Females who are pregnant or breastfeeding
* Concomitant receipt of any β-lactams antibiotic
* Concomitant receipt of probenecid
* Reduced kidney function defined as creatinine clearance of ≤ 50 mL/min
* Any other reason felt by the investigator to potentially affect the outcomes of the study

Experimental Group Only:

* No palpable pedal pulses present
* Participants likely to require multiple surgical interventions during the study period, which therefore could affect placement of the microdialysis catheter

Active Comparator Group Only:

* Positive urine drug screen (cocaine, tetrahydrocannabinol, opiates, benzodiazepines, and amphetamines)
* History of regular alcohol consumption exceeding 7 drinks/week for females or 14 drinks/week for men (1 drink = 5 ounces of wine or 12 ounces of beer or 1.5 ounces of hard liquor) within 6 months of screening.
* Use of tobacco- or nicotine-containing products in excess of the equivalence of 5 cigarettes per day.
* Use of prescription or nonprescription drugs, vitamins, or dietary supplements within 7 days or 5 half-lives (whichever is longer) prior to the first dose of study medication, with the exception of acetaminophen at doses of ≤ 1 g/day. Herbal supplements, hormonal methods of contraception (including oral and transdermal contraceptives, injectable progesterone, progestin subdermal implants, progesterone-releasing intrauterine devices (IUDs), postcoital contraceptive methods), and hormone replacement therapy must be discontinued at least 14 days prior to the first dose of study medication. Depo-Provera® must be discontinued at least 6 months prior to the first dose of study medication.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2016-02-19 (Actual); Primary Completion 2017-04 (Actual); Study Completion 2017-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David P Nicolau, PharmD, Principal Investigator — Harford Hospital
Locations (1):
- Hartford Hospital, Hartford, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Monogue ML, Stainton SM, Baummer-Carr A, Shepard AK, Nugent JF, Kuti JL, Nicolau DP. Pharmacokinetics and Tissue Penetration of Ceftolozane-Tazobactam in Diabetic Patients with Lower Limb Infections and Healthy Adult Volunteers. Antimicrob Agents Chemother. 2017 Nov 22;61(12):e01449-17. doi: 10.1128/AAC.01449-17. Print 2017 Dec. PMID 28893779

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Diabetic Wound Infection | Healthy Volunteer
Started | 10 | 6
Completed | 10 | 6
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Diabetic Wound Infection | Healthy Volunteer | Total
Number analyzed (Participants) | 10 | 6 | 16
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 1 | 1
  Between 18 and 65 years | 10 | 5 | 15
  >=65 years | 0 | 0 | 0
Age, Continuous [Median (Full Range); unit: years] | 53 [35 to 64] | 28 [18 to 36] | 44 [18 to 64]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 3
  Male | 9 | 4 | 13
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 10 | 6 | 16
Height [Median (Full Range); unit: centimeters] | 182.9 [164.0 to 193.0] | 170.2 [157.5 to 186.7] | 178.1 [157.5 to 193.0]
Weight [Median (Full Range); unit: kilograms] | 114.8 [74.6 to 147.0] | 69.1 [50.5 to 102.7] | 97.7 [50.5 to 147.0]
Body Mass Index [Median (Full Range); unit: kg/m^2] | 33.4 [26.6 to 48.0] | 24.0 [20.4 to 29.5] | 29.9 [20.4 to 48.0]
Creatinine clearance [Median (Full Range); unit: mL/min] | 108.4 [75.3 to 136.5] | 121.5 [92.5 to 159.2] | 113.3 [75.3 to 159.2]

OUTCOME MEASURES:

1. Primary Outcome: Ceftolozane Tissue Penetration
Description: The ratio of ceftolozane tissue concentration area under the curve (AUC) to plasma concentrations AUC following the final (i.e., 3rd) ceftolozane/tazobactam dose.
  Note. Ceftolozane/tazobactam doses were administered at 0, 8, and 16 hours. Plasma and dialysate concentrations were determined at hours 16, 17, 18, 19, 20, 21, 22, 23, and 24 hours after the first dose for determination of ceftolozane AUC in blood and tissue.
Time Frame: 16-24 hours
Measure: Median (Full Range); unit: ratio
Arm/Group | Diabetic Wound Infection | Healthy Volunteer
Number analyzed (Participants) | 10 | 6
ratio | 0.75 [0.35 to 1.00] | 0.87 [0.54 to 2.20]

2. Primary Outcome: Tazobactam Tissue Penetration
Description: The ratio of tazobactam tissue concentration area under the curve (AUC) to plasma concentration AUC following the final (3rd) ceftolozane/tazobactam dose.
  Note. Ceftolozane/tazobactam doses were administered at 0, 8, and 16 hours. Plasma and dialysate concentrations were determined at hours 16, 17, 18, 19, 20, 21, 22, 23, and 24 hours after the first dose for determination of tazobactam AUC in blood and tissue.
Time Frame: 16-24 hours
Population: Seven of the 10 enrolled participants in the Diabetic Wound Infection cohort provided data for tazobactam in plasma. Assay interference was observed in samples for two participants, and one participant had concentrations below the lower limit of the detection for the assay. This explains the difference with participant flow numbers.
Measure: Median (Full Range); unit: ratio
Arm/Group | Diabetic Wound Infection | Healthy Volunteer
Number analyzed (Participants) | 7 | 6
ratio | 1.18 [0.54 to 1.44] | 0.85 [0.63 to 2.10]

3. Secondary Outcome: Ceftolozane Area Under the Curve (AUC) in Tissue
Description: The ceftolozane AUC in tissue from 16 to 24 hours.
  Note. Ceftolozane/tazobactam doses were administered at 0, 8, and 16 hours. Dialysate concentrations were determined at hours 16, 17, 18, 19, 20, 21, 22, 23, and 24 hours after the first dose for determination of ceftolozane AUC.
Time Frame: 16 to 24 hours post-dose
Measure: Median (Full Range); unit: µg•h/mL
Arm/Group | Diabetic Wound Infection | Healthy Volunteer
Number analyzed (Participants) | 10 | 6
µg•h/mL | 121.5 [72.7 to 191.7] | 130.6 [95.4 to 189.4]

4. Secondary Outcome: Tazobactam AUC in Tissue
Description: The tazobactam AUC in tissue over 16 to 24 hours
  Note. Ceftolozane/tazobactam doses were administered at 0, 8, and 16 hours. Dialysate concentrations were determined at hours 16, 17, 18, 19, 20, 21, 22, 23, and 24 hours after the first dose for determination of tazobactam AUC.
Time Frame: 16 to 24 hours post-dose
Measure: Median (Full Range); unit: µg•h/mL
Arm/Group | Diabetic Wound Infection | Healthy Volunteer
Number analyzed (Participants) | 10 | 6
µg•h/mL | 15.8 [8.6 to 32.9] | 13.8 [7.7 to 18.7]

5. Secondary Outcome: Ceftolozane Total Drug AUC in Plasma
Description: The ceftolozane total drug AUC in plasma over 16 to 24 hours
  Note. Ceftolozane/tazobactam doses were administered at 0, 8, and 16 hours. Plasma concentrations were determined at hours 16, 17, 18, 19, 20, 21, 22, 23, and 24 hours after the first dose for determination of ceftolozane AUC.
Time Frame: 16 to 24 hours post-dose
Measure: Median (Full Range); unit: µg•h/mL
Arm/Group | Diabetic Wound Infection | Healthy Volunteer
Number analyzed (Participants) | 10 | 6
µg•h/mL | 191.6 [147.1 to 286.6] | 191.3 [118.1 to 274.3]

6. Secondary Outcome: Tazobactam Total Drug AUC in Plasma
Description: The tazobactam total drug AUC in plasma over 16 to 24 hours
  Note. Ceftolozane/tazobactam doses were administered at 0, 8, and 16 hours. Plasma concentrations were determined at hours 16, 17, 18, 19, 20, 21, 22, 23, and 24 hours after the first dose for determination of tazobactam AUC.
Time Frame: 16 to 24 hours post-dose
Population: as for outcome 2
Measure: Median (Full Range); unit: µg•h/mL
Arm/Group | Diabetic Wound Infection | Healthy Volunteer
Number analyzed (Participants) | 7 | 6
µg•h/mL | 27.1 [15.0 to 70.0] | 22.2 [19.2 to 36.4]

7. Secondary Outcome: Number of Participants With Adverse Events
Description: Number of reported or documented adverse events recorded during participation in the study.
Time Frame: Duration of study (34 hours)
Measure: Count of Participants; unit: Participants
Arm/Group | Diabetic Wound Infection | Healthy Volunteer
Number analyzed (Participants) | 10 | 6
Participants | 1 | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected until study completion (approximately 34 hours). All abnormal laboratory determinations were followed until resolution unless follow-up is determined to be unnecessary by the study physician. For the control group, participants were discharged from the study after a 4 hour monitoring period from removal of microdialysis catheters.
Description: Adverse event: any pathologic or unintended change in the structure, function, or chemistry associated with the use of the study drug, whether or not considered drug related:
  MILD - present, but easily tolerated MODERATE - discomfort that interferes with usual activities SEVERE - incapacitating, inability to do usual activities A serious adverse event will be defined as any which results in death or is immediately life-threatening, requires in-participant hospitalization.
Arm/Group | Diabetic Wound Infection | Healthy Volunteer
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/6
Other Adverse Events (participants affected / at risk) | 1/10 | 0/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Diabetic Wound Infection (N=10) | Healthy Volunteer (N=6)
Vertigo (Nervous system disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
No clinical or microbiological outcome data were collected; patient and volunteers were not matched based on demographic data; interference with the plasma assay was observed in two patients.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-06-27): https://cdn.clinicaltrials.gov/large-docs/74/NCT02620774/Prot_SAP_000.pdf